CLINICAL TRIAL: NCT05790161
Title: Consequences of Caffeine Intake in Teenagers: Effects on Sleep, Reward Processing, Risk Taking, and Underlying Cerebral Mechanisms Under Conditions of Sleep Restriction
Brief Title: Consequences of Caffeine Intake in Sleep Restricted Teenagers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Psychiatric Hospital of the University of Basel (Other)
Collaborators: University of Zurich (Other); University of Basel (Other); University Hospital, Basel, Switzerland (Other); University of Pittsburgh (Other); University of Liege (Other)
Responsible Party: Principal Investigator, Carolin Reichert, Deputy Head, Psychiatric Hospital of the University of Basel
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CaReTeens
Record Dates: First submitted 2023-03-04; First posted 2023-03-30 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Caffeine; Insufficient Sleep
Keywords: adolescence; sleep; caffeine; Risk-Taking; reward
MeSH Terms: conditions — Sleep Deprivation; Risk-Taking | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: Within-Design regarding treatment (caffeine vs. placebo). Between-Design regarding sleep manipulation (sleep restriction vs. sleep manipulation)
Who Masked: Participant, Investigator
Masking Description: doubleblind regarding treatment no blinding regarding sleep manipulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Restriction (Experimental): 3 nights with 6h sleep opportunity each.
  Interventions: Drug: Caffeine
- Sleep Extension (Experimental): 3 nights with 9,5h sleep opportunity each.
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — 2mg/kg, once before night 6 and once before the scan (either on week 1 or 2, alternating with placebo)

SUMMARY:
The goal of this clinical trial is to systematically investigate two prominent factors in teenagers' daily life: Caffeine and sleep restriction (SR) and their combined influence on sleep, cognition, and behavior in healthy adolescents. The main questions it aims to answer are:

The effects of caffeine under conditions of SR and SE:

* on sleep pressure and sleep continuity.
* on BOLD activity differences in reward related areas during a reward task (monetary incentive delay task) and on reaction times (behavioral aspect) in the same task.
* on BOLD activity differences during a risk taking task (wheel of fortune task) and on risky decision-making (behavioral aspect) in the same task.

Participants will be either in the SR or SE condition (between-subject). The protocol consists of 2x of approximately one week in which a participant will receive caffeine or placebo (within-subject) at the last two evenings.

The experiment consists of an ambulatory and a laboratory phase:

* The ambulatory phase consists of 5 nights, including 3 stabilization nights (8h sleep opportunity) prior to 2 nights consisting of either SR with 6h sleep opportunity or SE with 9.5h sleep opportunity. Participants will wear an actiwatch and fill out sleep diaries during this period.
* The laboratory phase will be the 6th evening, night and morning of the protocol and will be spent in our lab. Participants will do the following:
* treatment (caffeine vs. placebo) intake
* saliva sampling
* drug screening
* cognitive tests, including risk-taking and reward task
* filling in questionnaires (sleep diary, sleep quality, sleepiness, mood, expectancy)
* waking and sleep with EEG

The next day, participants will undergo an fMRI scan, including the following:

* resting-state scan
* structural scan
* arterial spin labeling scan
* reward task scan
* risk-taking task scan

Around the scan, participants will fill out/undergo:

* saliva sampling
* questionnaires (reward task, mood, sleepiness, expectancy)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 14 and ≤ 17
* Clinically healthy
* Signed consent form of participant and legal guardian

Exclusion Criteria:

* Inability to operate tasks or understand the study information
* Participation in other clinical trials <3 months prior to any possible study start date
* BMI P3 < BMI-PC < P97
* Any general health concerns or disorders (previous diagnosis of heart/cardiovascular/nephrological/endocrinological/diabetic/metabolic/chronobiologic/ psychiatric/neurological [particularly epilepsy and parasomnia] conditions) which may make participants vulnerable to potential negative effects of SR or caffeine or which may affect outcome measures
* Unavailability to complete the two study protocol weeks within a three-month period
* Trans meridian travel (>2 time zones) <1 month before any possible study start date
* Shift work <3 months prior to any possible study start date
* Extreme chronotype MSFSC < 3:00 / MSFSC > 6:00 according to MCTQ
* Subjective sleep duration on school days <7h or >9h according to MCTQ
* Metallic prosthesis, metallic implants, or non-removable objects in the body (e.g., splinters, piercings) which affect MRI safety
* Tattoos with larger diameter than 10cm or above shoulder area, affecting MRI safety
* Claustrophobia
* Difficulties or problems in physical well-being and mental health based on the Swiss norm (T< 35) for all genders aged 12-18 according to KIDSCREEN-27
* Daily nicotine use
* Use of medications or drugs that have contraindications and/or effects on outcome measures or use of specific drugs indicated in drug test
* Use of alcohol to an extent that it is likely to have contraindications and/or effects on outcome measures
* Any indication of previous withdrawal or oversensitivity to caffeine
* Sleep quality >5 according to PSQI
* Problems of EEG compatibility
* Sleep efficiency <70%
* Identification of sleep disorders
* Pregnancy
* Deviation from the stabilisation sleep-wake schedule by +-60 mins
* Deviation from protocol sleep-wake schedule by +-30 mins

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Nighttime Sleep SWA | Laboratory night week 1
  Sleep at night will be quantified by polysomnographic recordings. Data will be scored epoch by epoch according to standard criteria to assign sleep stages. Spectral analysis will be performed by applying fast Fourier transformation. The key marker of sleep pressure will be slow wave activity (SWA) during NREM sleep (i.e., stage 2+3) defined as EEG power density between 0.75-4.5 Hz. To specify potential effects on SWA more precisely the investigators will additionally conduct separate analyses within this band and with separate (0.5 Hz) bins. To characterize the effects of the experimental manipulation on sleep more comprehensively, the investigators will also conduct analyses on different time bins within one night (e.g. time bin of the first 5 hours of sleep), and on different sleep stages (including wakefulness and latency to sleep), and bands other than SWA. If our resources allow, the investigators will also explore the effects of our experimental manipulation on slow wave energy.
Nighttime Sleep SWA | Laboratory night week 2
  Sleep at night will be quantified by polysomnographic recordings. Data will be scored epoch by epoch according to standard criteria to assign sleep stages. Spectral analysis will be performed by applying fast Fourier transformation. The key marker of sleep pressure will be slow wave activity (SWA) during NREM sleep (i.e., stage 2+3) defined as EEG power density between 0.75-4.5 Hz. To specify potential effects on SWA more precisely the investigators will additionally conduct separate analyses within this band and with separate (0.5 Hz) bins. To characterize the effects of the experimental manipulation on sleep more comprehensively, the investigators will also conduct analyses on different time bins within one night (e.g. time bin of the first 5 hours of sleep), and on different sleep stages (including wakefulness and latency to sleep), and bands other than SWA. If our resources allow, the investigators will also explore the effects of our experimental manipulation on slow wave energy.
BOLD activity during reward processing | fMRI session week 1
  BOLD activity will be measured with a 3T MRT scanner. Brain responses will be modeled in an event-related design using a GLM for each subject at each voxel/trial. Regressors of no interest include motion parameters & amount of gain or loss. At a within-subject level, the investigators contrast BOLD activity in caffeine vs placebo conditions (& vice versa). The investigators focus on BOLD activity differences in reward-related regions between anticipation of reward vs neutral events. At the random effects level, the investigators test for the effects of SR vs SE (& vice versa) and the interaction with caffeine vs placebo. The investigators report whole-brain results. Corrections for multiple comparisons will be made accordingly. The investigators measure RTs to expected rewards, losses, and neutral trials. Task difficulty is individually adapted throughout the task.
BOLD activity during reward processing | fMRI session week 2
  BOLD activity will be measured with a 3T MRT scanner. Brain responses will be modeled in an event-related design using a GLM for each subject at each voxel/trial. Regressors of no interest include motion parameters & amount of gain or loss. At a within-subject level, the investigators contrast BOLD activity in caffeine vs placebo conditions (& vice versa). The investigators focus on BOLD activity differences in reward-related regions between anticipation of reward vs neutral events. At the random effects level, the investigators test for the effects of SR vs SE (& vice versa) and the interaction with caffeine vs placebo. The investigators report whole-brain results. Corrections for multiple comparisons will be made accordingly. The investigators measure RTs to expected rewards, losses, and neutral trials. Task difficulty is individually adapted throughout the task.
BOLD activity during risk-decision making (RDM) | fMRI session week 1
  BOLD activity/brain responses will be measured as above. Regressors of no interest additionally include risk probability, indicated amount of gain & difference in expected value between safe and risky option. At within-subject level, the investigators contrast BOLD activity in caffeine vs placebo conditions (&vice versa). If number of events is sufficient, the investigators focus on BOLD activity differences in regions related to RDM between safe/risky choices. At the random effects level, the investigators test for effects of SR vs SE (&vice versa) & the interaction with caffeine vs placebo. The investigators report whole-brain results Connectivity analyses to characterize brain activity underlying RDM are planned.
BOLD activity during risk-decision making (RDM) | fMRI session week 2
  BOLD activity/brain responses will be measured as above. Regressors of no interest additionally include risk probability, indicated amount of gain & difference in expected value between safe and risky option. At within-subject level, the investigators contrast BOLD activity in caffeine vs placebo conditions (&vice versa). If number of events is sufficient, the investigators focus on BOLD activity differences in regions related to RDM between safe/risky choices. At the random effects level, the investigators test for effects of SR vs SE (&vice versa) & the interaction with caffeine vs placebo. The investigators report whole-brain results Connectivity analyses to characterize brain activity underlying RDM are planned.

SECONDARY OUTCOMES:
Resting state(rs) functional connectivity (FC) | fMRI session week 1; fMRI session week 2
  Rs-FC will be ascertained via BOLD measured with MRI in a 3T Siemens scanner (Prisma; Siemens AG, Erlangen, Germany) using a 24-channel head coil. The standard three-dimensional magnetization-prepared rapid acquisition (MPRAGE) sequence with gradient echo (1x1x1mm, TR=2000ms, TI= 1000ms, TE=3.37ms, FA=8°) will obtain T1-weighted images to depict morphological aspects of the brain. To depict BOLD activity during resting T2*-weighted echo-planar image (EPI) sequences (TR = 2000, TE = 35ms, FOV = 216mm, voxel size = 2.4 mm3, matrix size 90*90, 50 slices) will be performed twice for 6-minutes. Foam and inflatable pads will be used to reduce head motion. Participants will be required to have eyes open and stare at a fixation cross to provide greater reliability of within-network connections and reduce experimental variability. Heart rate and respiration will be recorded by Siemens MRI scanner installed hardware.
BOLD activity during reward feedback | fMRI session week 1; fMRI session week 2
  BOLD activity will be measured with a 3T MRT scanner. Brain responses will first be modeled in an event-related design using a GLM for each subject at each voxel and each trial. Regressors of no interest include motion parameters and indicated amount of gain or loss (high vs low) and the type of feedback. At a within-subject level, the investigators contrast BOLD activity in caffeine vs placebo (and vice versa). The investigators focus on differences in reward-related regions between feedback of successful reward trials vs successful neutral trials. The investigators may run analyses contrasting feedback of successful reward trials vs feedback of neutral trials. At the 2nd (random effects) level, the investigators test for effects of SR vs SE (and vice versa) and interaction with caffeine vs placebo. The investigators correct for multiple comparisons within reward-related regions. The investigators report whole-brain results, corrected for whole brain multiple comparisons.
Vigilance | Laboratory evening (3 times) and morning (1 time SE & 2 times SR) week 1; Laboratory evening (3 times) and morning (1 time SE & 2 times SR) week 2
  Vigilance performance will be quantified by mean 1/RT for all reaction times in the Psychometric Vigilance Task. The investigators may also report the number of lapses (trials with RT > 500ms) if meaningful and may explore the effects of our experimental manipulation on other typical outcome variables of the PVT.
Working Memory | LaboratoryLaboratory evening (1 time) and morning (1 time) week 1; Laboratory evening (1 time) and morning (1 time) week 2
  Working Memory will be quantified by RT, number of n-back reached, and accuracy (number of missings, number of hits) in an adaptive n-back task. The n-back task is a computer-based task to assess working memory performance. The participant is presented with a sequence of stimuli and must indicate when the current stimulus matches the one from n steps earlier in the sequence. The investigators will use an adaptive n-back version where the n steps adapt to individual performance
Inihibition | Laboratory evening (2 times) and morning (1 time SE & 2 times SR) week 1; Laboratory evening (2 times) and morning (1 time SE & 2 times SR) week 2
  Inhibition performance will be quantified by the number of commission and omission errors in a go/nogo task. The investigators will also report RTs. The participants will be asked to press a button in response to visually presented stimuli, but to avoid responding to a rarer nontarget.
Subjective Sleepiness | Laboratory evening (7 times) and morning (2 times SE & 4 times SR ) week 1; Laboratory evening (7 times) and morning (2 times SE & 4 times SR ) week 2
  Subjective sleepiness will be quantified by the Karolinska Sleepiness Scale (KSS). This is a 9-point scale (1 = extremely, alert, 3 = alert, 5 = neither alert nor sleepy, 7 = sleepy - but no difficulty remaining awake, and 9 = extremely sleepy - fighting sleep) which the participants are asked to fill in.
Circadian timing (DLMO) | laboratory phase week 1 (9 samples SE & 11 samples SR) & fMRI Session week 1 (3 samples) ;laboratory phase week 2 (9 samples SE & 11 samples SR) & fMRI Session week 2 (3 samples)
  The investigators will measure melatonin levels in saliva samples using biochemical analysis. The investigators will report melatonin levels and melatonin suppression. Dim-light melatonin onset (DLMO) will be the indicator for the onset of the biological night and quantified using the hockey-stick method.
Objective Sleepiness | Laboratory evening (3 times) and morning (1 time SE & 2 times SR) week 1; Laboratory evening (2 times) and morning (1 time) week 2
  The investigators will quantify sleepiness objectively via EEG delta and theta activity (ranges ~0.5-8 Hz) in a 3-minute Waking-EEG where participants will be asked to stare at a fixation cross or during task performance.
Subjective Sleep Quality | Laboratory morning week 1 (1 time); Laboratory morning (1 time) week 2
  To measure subjective sleep quality, the investigators use the Leeds Sleep Evaluation Questionnaire (LSEQ) administered in the morning after wake-up. The questionnaire results in values on the four dimensions: Getting to Sleep, Quality of Sleep, Awake Following Sleep, and Behaviour Following Wakening.

CONTACTS AND LOCATIONS:
Overall Officials: Carolin Reichert, Dr., Principal Investigator — University of Basel
Locations (1):
- Centre for Chronobiology, Basel, Switzerland